CLINICAL TRIAL: NCT06313242
Title: Evaluation of Different Bowel Preparations in Magnetically Controlled Capsule Endoscopy: a Randomized Controlled Study
Brief Title: Different Bowel Preparations in Magnetically Controlled Capsule Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202403
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Magnetically Controlled Capsule Endoscopy; Bowel Preparation
MeSH Terms: interventions — Laxatives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laxatives arm (Active Comparator): Normal diet 1 day before the test, fasting and laxatives from 20:00 pm. The laxatives, Polyethylene Glycol Electrolytes Powder (II), should be prepared as a solution and taken as 2000 ml the night before the test and 1000 ml the following morning, within 2 hours and 1 hour, respectively.
  Interventions: Drug: Polyethylene Glycol Electrolytes Powder (II)
- Low residue diet arm (Experimental): Low residue diet 1 day before the test, fasting from 20:00 pm.
  Interventions: Other: Low residue diet
- Normal diet arm (Experimental): Normal diet 1 day before the test, fasting from 20:00 pm.
  Interventions: Other: Normal diet

INTERVENTIONS:
Drug: Polyethylene Glycol Electrolytes Powder (II) — Polyethylene Glycol Electrolytes Powder (II) was used for bowel preparation.
  Other Names: laxatives for bowel preparation
  Arms: Laxatives arm
Other: Low residue diet — Low residue diet 1 day before the test, fasting from 20:00 pm.
  Arms: Low residue diet arm
Other: Normal diet — Normal diet 1 day before the test, fasting from 20:00 pm.
  Arms: Normal diet arm

SUMMARY:
The study aimed to compare the effects of bowel preparation methods of a normal diet for 1 day, a low residue diet for 1 day, and laxative bowel cleaning on the image quality of magnetically controlled capsule endoscopy, and to assess the rate of completion of the examination, small intestine transit time, lesion detection, patient tolerance, and safety of the three regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female
2. One of the following examination indications:

(1) Unexplained gastrointestinal bleeding; (2) Unexplained iron deficiency anaemia; (3) Suspected Crohn's disease or monitoring and directing treatment for Crohn's disease; (4) Suspected small bowel tumour; (5) Monitoring the development of small bowel polyposis syndrome; (6) Suspected or difficult to control malabsorption syndromes (e.g., celiac disease, etc.); (7) Detection of NSAID-associated small bowel mucosal damage; (8) Those with a clinical need to exclude small bowel disease.

Exclusion Criteria:

1. People who are ineligible for surgery or refuse to undergo any abdominal surgery (once the capsule is retained it cannot be removed surgically);
2. Known or suspected gastrointestinal obstruction, stenosis, and fistula;
3. People with implanted cardiac pacemakers or other electronic devices;
4. People with swallowing disorders;
5. Women during pregnancy;
6. People who are unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Image quality of small intestine | 1 day (Upon completion of the examination)
  The small bowel cleanliness score and the small bowel bubble volume score were used to evaluate image quality.

SECONDARY OUTCOMES:
Rate of completion of inspections | 1 day (Upon completion of the examination)
  The examination is considered complete when the capsule reaches the cecum.
Small intestine transit time | 1 day (Upon completion of the examination)
  Time taken for the capsule to pass through the entire small intestine to reach the cecum.
Lesion detection rate | 1 day (Upon completion of the examination)
  Proportion of cases with lesions relevant to the indication for examination or capable of explaining the patient's complaints or symptoms to the total number of cases.
Patient tolerance | 1 day (Upon completion of the examination)
  Evaluated by completing a case report form based on the patient's personal feelings during the bowel preparation process.
Rate of adverse events | 1 day (Upon completion of the examination)
  Patients were observed for adverse events (nausea, vomiting, bloating, etc.) and for capsule retention after examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han Y, Liao Z, Li Y, Zhao X, Ma S, Bao D, Qiu M, Deng J, Wang J, Qu P, Jiang C, Jia S, Yang S, Ru L, Feng J, Gao W, Huang Y, Tao L, Han Y, Yang K, Wang X, Zhang W, Wang B, Li Y, Yang Y, Li J, Sheng J, Ma Y, Cui M, Ma S, Wang X, Li Z, Stone GW. Magnetically Controlled Capsule Endoscopy for Assessment of Antiplatelet Therapy-Induced Gastrointestinal Injury. J Am Coll Cardiol. 2022 Jan 18;79(2):116-128. doi: 10.1016/j.jacc.2021.10.028. Epub 2021 Nov 6. PMID 34752902
- [Background] Wu TT, Zhang MY, Tan ND, Chen SF, Zhuang QJ, Luo Y, Xiao YL. Patients at risk for further examination with conventional gastroscopy after undergoing magnetically controlled capsule endoscopy. J Dig Dis. 2023 Oct;24(10):522-529. doi: 10.1111/1751-2980.13228. Epub 2023 Oct 3. PMID 37681236
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Kong QZ, Peng C, Li Z, Tian BL, Li YY, Chen FX, Zuo XL, Li YQ. Inadequate gastric preparation and its associated factors for magnetically controlled capsule endoscopy. Front Pharmacol. 2023 Aug 28;14:1184754. doi: 10.3389/fphar.2023.1184754. eCollection 2023. PMID 37701026
- [Background] Reumkens A, van der Zander Q, Winkens B, Bogie R, Bakker CM, Sanduleanu S, Masclee AAM. Electrolyte disturbances after bowel preparation for colonoscopy: Systematic review and meta-analysis. Dig Endosc. 2022 Jul;34(5):913-926. doi: 10.1111/den.14237. Epub 2022 Feb 23. PMID 35037327
- [Background] Gkolfakis P, Tziatzios G, Dimitriadis GD, Triantafyllou K. Meta-analysis of randomized controlled trials challenging the usefulness of purgative preparation before small-bowel video capsule endoscopy. Endoscopy. 2018 Jul;50(7):671-683. doi: 10.1055/s-0043-125207. Epub 2018 Feb 6. PMID 29409067
- [Background] Gomez-Reyes E, Tepox-Padron A, Cano-Manrique G, Vilchis-Valadez NJ, Mora-Bulnes S, Medrano-Duarte G, Chaires-Garza LG, Grajales-Figueroa G, Ruiz-Romero D, Tellez-Avila FI. A low-residue diet before colonoscopy tends to improve tolerability by patients with no differences in preparation quality: a randomized trial. Surg Endosc. 2020 Jul;34(7):3037-3042. doi: 10.1007/s00464-019-07100-6. Epub 2019 Sep 3. PMID 31482360
- [Background] Nguyen DL, Jamal MM, Nguyen ET, Puli SR, Bechtold ML. Low-residue versus clear liquid diet before colonoscopy: a meta-analysis of randomized, controlled trials. Gastrointest Endosc. 2016 Mar;83(3):499-507.e1. doi: 10.1016/j.gie.2015.09.045. Epub 2015 Oct 13. PMID 26460222